CLINICAL TRIAL: NCT05965752
Title: RECOVER-NEURO: A Platform Protocol for Evaluation of Interventions for Cognitive Dysfunction in Post-Acute Sequelae of SARS-CoV-2 Infection (PASC)
Brief Title: RECOVER-NEURO: Platform Protocol to Measure the Effects of Cognitive Dysfunction Interventions on Long COVID Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00112477; OTA-21-015G (Other Grant/Funding Number: NIH grant to RTI; RTI subcontracting with DCRI)
Record Dates: First submitted 2023-07-25; First posted 2023-07-28 (Actual); Results first posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Long COVID; Long COVID-19; Long COVID19
Keywords: PASC; Cognitive
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: To achieve blinding and an equitable randomization probability, a two-step randomization process will be used. The study will employ a simple (unstratified) randomization scheme.
  At the first stage, each participant will be assigned with equal probability to one of the intervention appendices for which the participant is eligible, after applying any intervention-specific safety exclusions. At the second stage, each participant will be assigned according to the specific appendix's randomization procedure. Participants will have an equal chance of being randomized into any of the intervention groups.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants assigned to active comparator will be considered part of pooled analyses if the intervention was active at the time of the participant's enrollment and the participants were eligible to receive that intervention. This will result in approximately a 1:1 allocation ratio for any intervention to pooled control.
  Sites will be informed to which intervention appendix participants are randomized, but, when applicable, not whether the participants are allocated to the active intervention arm or active comparator arm within that appendix. The participants and investigators will be blinded throughout the study, when possible.
  If open intervention appendices do not have the ability to pool controls but have independent controls, at the second stage participants will be randomized in a 1:1 ratio to intervention vs active comparator inside the specific intervention appendix the participants were randomized to at the first stage of the randomization procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- BrainHQ Active Comparator (Active Comparator): 5 sessions/week at 30 min/session
  Interventions: Other: BrainHQ/Active Comparator Activity
- BrainHQ (Experimental): 5 sessions/week at 30 min/session
  Interventions: Other: BrainHQ
- BrainHQ + PASC CoRE (Experimental): BrainHQ plus 9 group sessions at 1.5 hr/session and 3 individual sessions at 30 min/session
  Interventions: Other: BrainHQ; Other: PASC CoRE
- Brain HQ + tDCS-active (Experimental): 2.0 mA stimulation delivered for 30 min during each BrainHQ session
  Interventions: Other: BrainHQ; Device: tDCS-active
- Brain HQ + tDCS-sham (Placebo Comparator): Inactive stimulation delivered for 30 min during each BrainHQ session
  Interventions: Other: BrainHQ; Device: tDCS-sham

INTERVENTIONS:
Other: BrainHQ/Active Comparator Activity — BrainHQ platform provides a set of cognitive activities, like puzzles and games, that are cognitively stimulating and actively engage participants but do not continuously and adaptively challenge them. These activities are designed to be a face-valid, active comparison approach to cognitive therapy, thus participants are blinded, attention time is matched, and overall user experience is identical to the active arms.
  Arms: BrainHQ Active Comparator
Other: BrainHQ — BrainHQ is an online cognitive training program, and has been used to improve cognitive function among persons with cognitive impairment based on principles of neuroplasticity.
  Arms: Brain HQ + tDCS-active; Brain HQ + tDCS-sham; BrainHQ; BrainHQ + PASC CoRE
Other: PASC CoRE — PASC CoRE is a manualized, adaptable cognitive rehabilitation intervention adapted from Goal Management Training and other evidence based programs that improve attention and executive functions, among other cognitive domains.
  Arms: BrainHQ + PASC CoRE
Device: tDCS-active — Transcranial direct current stimulation (tDCS) will use a device specifically for home-based use. This device delivers a weak electrical current of 2.0 mA passed through two electrodes placed on the scalp to target the dorsolateral prefrontal cortex region of the brain. The electrodes are single-use for each session and can be attached to a headset by snapping into place.
  The device has a user-friendly interface and a large-button keypad, making it is easy to use at home.
  Arms: Brain HQ + tDCS-active
Device: tDCS-sham — tDCS devices used in the sham arm will be pre-programmed to deliver the same ramp up/down at the beginning/end of the 30-minute period as the active arm, except with no current otherwise delivered during the session.
  Arms: Brain HQ + tDCS-sham

SUMMARY:
This platform protocol is designed to be flexible so that it is suitable for a wide range of settings within health care systems, for remote settings, and in community settings where it can be integrated into COVID-19 programs and subsequent treatment plans.

This protocol is a prospective, multi-center, multi-arm, randomized, controlled platform trial evaluating potential interventions for PASC-mediated cognitive dysfunction. The hypothesis is that PASC associated dysfunction in cognitive domains, such as executive function and attention, may be improved by interventions that selectively focus on enhancing those domains.

DETAILED DESCRIPTION:
Participants will be randomized to one of the intervention appendices that are actively enrolling at the time of randomization. Intervention appendices may be added or removed according to adaptive design and/or emerging evidence. Various interventions will be studied.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. ≥ 18 years of age at the time of enrollment
2. PROMIS-Cog T-score < 40
3. Previous suspected, probable, or confirmed SARS-CoV-2 infection, as defined by the Pan American Health Organization

   Suspected case of SARS-CoV-2 infection - three options, A through C:

   A. Met clinical OR epidemiological criteria:

   a. Clinical criteria: Acute onset of fever AND cough (influenza-like illness) OR Acute onset of ANY THREE OR MORE of the following signs or symptoms: fever, cough, general, weakness/fatigue, headache, myalgia, sore throat, coryza, dyspnea, nausea, diarrhea, anorexia; b. Epidemiological criteria: Contact of a probable or confirmed case or linked to a COVID-19 cluster;

   B. Presented acute respiratory infection with history of fever or measured fever of ≥ 38°C and cough, with onset within the last 10 days, and who requires hospitalization; or

   C. Presented with no clinical signs or symptoms, NOR meeting epidemiologic criteria with a positive professional use or self-test SARS-CoV-2 Antigen-Rapid Diagnostic Test.

   Probable case of SARS-CoV-2 infection, defined as having met clinical criteria above AND was a contact of a probable or confirmed case or was linked to a COVID-19 cluster.

   Confirmed case of SARS-CoV-2 infection - two options, A through B:

   A. Presented with a positive nucleic acid amplification test, regardless of clinical criteria OR epidemiological criteria; or

   B. Met clinical AND/OR epidemiological criteria (See suspected case A.a.), with a positive professional use or self-test SARS-CoV-2 Antigen-Rapid Diagnostic Test.

   * Suspected and probable cases will only be allowed if they occurred before May 1, 2021, and will be limited to 10% of the study population. Otherwise, confirmed cases are required.
4. Cognitive dysfunction symptoms following a SARS-CoV-2 infection that have persisted for at least 12 weeks and are still present at the time of consent
5. Fluent in English or Spanish language
6. Willing and able to provide informed consent, complete the intervention, complete the intervention assessments, and return for all of the necessary follow-up visits

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Prior or active unstable or progressive major psychiatric or neurologic condition that would not show improvement and could hide treatment effect and is not related to SARS-CoV-2 infection, at the investigator's discretion, including, but not limited to, the following examples:

   a. Progressive neurodegenerative disease, such as Alzheimer's disease, Parkinson's disease, etc.

   b. Past traumatic brain injury occurrence still associated with active post-concussive symptoms c. Uncontrolled seizure disorder, such as having at least one seizure in the last year that is adjudicated by clinical judgement d. Post-stroke deficits that may interfere with assessment, such as language or communication difficulties, aphasia, etc.

   e. Formal thought disorders, such as schizophrenia, etc. f. Any neuropsychiatric or neurologic disorder uncontrolled for the previous six months or that may interfere with assessment, at discretion of the investigator
2. Known prior diagnosis of myalgic encephalomyelitis/chronic fatigue syndrome, not related to SARS-CoV-2 infection
3. Known active acute SARS-CoV-2 infection ≤ 4 weeks from consent
4. Current use of symptomatic therapies including prescribed or illicit stimulants, amantadine, N-methyl-D-aspartate receptor antagonists (e.g., memantine, dissociative drugs)
5. Current use of a stimulant for treating any PASC-related symptom
6. Current diagnosis of alcohol and substance use disorders

   a. Prior use disorders acceptable if abstinence achieved and maintained for at least 12 months before study enrollment
7. Insufficient visual, auditory, and motor function to participate in intervention and assessments
8. Known pregnancy
9. Current or recent use (within the last 2 months) of intervention*
10. Known allergy/sensitivity/hypersensitivity to components of the intervention or comparator*
11. Currently receiving/using intervention from another clinical trial, such as another RECOVER trial
12. Any condition that would make the participant, in the opinion of the investigator, unsuitable for the study

    1. The site investigator has the discretion to determine whether a participant is too cognitively impaired to participate and should instead be referred for clinical evaluation.

Exclusions specific to intervention appendices are listed in each appendix.

* Relevant if only one intervention appendix is open at the time of enrollment, though exclusion may be qualified in the appendix. If multiple intervention appendices are open, a participant may be excluded from any intervention appendix based on contraindications listed in the intervention appendix, current use of intervention, or known allergy/sensitivity/hypersensitivity and still remain eligible for the remaining intervention appendices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kanecia Zimmerman, MD PhD, Study Chair — Duke University; Daniel Laskowitz, MD MHS, Study Chair — Duke University
Locations (24):
- United States (24):
  - Banner University Medical Center Phoenix, Phoenix, Arizona
  - Banner University Medical Center- Tucson, Tucson, Arizona
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Stanford University, Stanford, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Florida College of Medicine Jacksonville, Jacksonville, Florida
  - Rush University Medical Center, Chicago, Illinois
  - OSF Healthcare, Peoria, Illinois
  - North Shore University Health System/Evanston Hospital, Skokie, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Jadestone Clinical Research, Silver Spring, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Daeconess Medical Center, Boston, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - NYU Langone Health/Brooklyn Hospital, Brooklyn, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Case Western Reserve University, Cleveland, Ohio
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Utah Hospitals and Clinics, Salt Lake City, Utah
  - University of Vermont, Burlington, Vermont
  - University of Washington, Seattle, Washington
  - West Virginia Clinical and Translational Science Institute, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No
The investigators will share the summary of results on the study website: https://recovercovid.org/

REFERENCES:
- See also: Related Info — http://recovercovid.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Brain HQ + tDCS-active: 2.0 mA stimulation delivered for 30 min during each BrainHQ session
  BrainHQ: BrainHQ is an online cognitive training program, and has been used to improve cognitive function among persons with cognitive impairment based on principles of neuroplasticity.
  tDCS-active: Transcranial direct current stimulation (tDCS) will use a device specifically for home-based use. This device delivers a weak electrical current of 2.0 mA passed through two electrodes placed on the scalp to target the dorsolateral prefrontal cortex region of the brain. The electrodes are single-use for each session and can be attached to a headset by snapping into place.
  The device has a user-friendly interface and a large-button keypad, making it is easy to use at home.
Period: Overall Study
Arm/Group | BrainHQ Active Comparator | BrainHQ | BrainHQ + PASC CoRE | Brain HQ + tDCS-active | Brain HQ + tDCS-sham
Started | 64 | 67 | 66 | 66 | 65
Completed | 59 | 62 | 62 | 55 | 58
Not Completed | 5 | 5 | 4 | 11 | 7
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 3
Not completed — Lost to Follow-up | 2 | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 1 | 5 | 0
Not completed — Disease Relapse | 1 | 0 | 1 | 0 | 0
Not completed — Failure to Meet Randomization Criteria | 0 | 1 | 0 | 1 | 0
Not completed — Unable to Return for Study Visits | 0 | 1 | 0 | 3 | 1
Not completed — Early Termination | 0 | 0 | 1 | 0 | 0
Not completed — Reported Unwanted Symptoms | 0 | 0 | 0 | 0 | 1
Not completed — Did Not Want to be Randomized to Intervention | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BrainHQ Active Comparator | BrainHQ | BrainHQ + PASC CoRE | Brain HQ + tDCS-active | Brain HQ + tDCS-sham | Total
Number analyzed (Participants) | 64 | 67 | 66 | 66 | 65 | 328
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 44.5 [37.5 to 55.0] | 49.0 [36.0 to 59.0] | 53.0 [41.0 to 58.0] | 47.0 [37.0 to 58.0] | 49.0 [35.0 to 57.0] | 48.0 [37.0 to 58.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 49 | 49 | 46 | 45 | 241
  Male | 12 | 18 | 17 | 20 | 20 | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 12 | 9 | 11 | 14 | 52
  Not Hispanic or Latino | 57 | 55 | 56 | 55 | 51 | 274
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 1 | 0 | 0 | 4
  Asian | 2 | 2 | 6 | 2 | 3 | 15
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 6 | 12 | 7 | 10 | 12 | 47
  White | 47 | 46 | 49 | 50 | 43 | 235
  More than one race | 5 | 3 | 2 | 3 | 2 | 15
  Unknown or Not Reported | 2 | 2 | 1 | 1 | 5 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 64 | 67 | 66 | 66 | 65 | 328

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Participants Enrolled in Each Appendix
Description: Appendix-specific outcome measure data will be reported under the associated NCT ID.
Time Frame: 160 Days
Population: Enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | BrainHQ Active Comparator | BrainHQ | BrainHQ + PASC CoRE | Brain HQ + tDCS-active | Brain HQ + tDCS-sham
Number analyzed (Participants) | 64 | 67 | 66 | 66 | 65
Participants | 64 | 67 | 66 | 66 | 65

ADVERSE EVENTS:
Time Frame: Up to approximately 160 days
Description: All-cause mortality events were collected during screening and from start of intervention to end of intervention. SAEs (Serious Adverse Events) and non-serious AEs were only collected from start of intervention to end of intervention and will be reported under each associated appendix's NCT ID.
Arm/Group | BrainHQ Active Comparator | BrainHQ | BrainHQ + PASC CoRE | Brain HQ + tDCS-active | Brain HQ + tDCS-sham
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/67 | 0/66 | 0/66 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-10): https://cdn.clinicaltrials.gov/large-docs/52/NCT05965752/Prot_SAP_001.pdf
  • Informed Consent Form (2024-02-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT05965752/ICF_000.pdf